CLINICAL TRIAL: NCT06147557
Title: Effect of Repeated Brief Passive Heat Therapy on Metabolism in Healthy Young Adults
Brief Title: Effect of Passive Heat Therapy on Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LithuananianSportsU-16
Record Dates: First submitted 2023-11-15; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat therapy (Experimental): 14 heat sessions of whole-body immersed in a 45°C water bath for 5 minutes.
  Interventions: Procedure: Heat therapy

INTERVENTIONS:
Procedure: Heat therapy — 14 heat sessions, during each session subjects were fully immersed in a 45°C water bath for 5 minutes.

SUMMARY:
The goal of this prospective interventional study is to examine if repeated brief hot stimuli affects glucose metabolism and substrate oxidation in young non-obese adults. Young adult participants were asked to participate in fourteen 5-min procedures involving whole body passive heating at 45°C water.

The main question it aims to answer is: "Does repeated brief noxious heat stimuli is sufficient to improve glucose tolerance, insulin sensitivity, and fat oxidation in young non-obese adults?"

DETAILED DESCRIPTION:
No studies yet addressed whether brief heat stimuli could be viable time-efficient alternative approach in order to improve glucose metabolism and fat oxidation. Consequently, we aimed to examine the ability of brief noxious heat stimuli to improve glucose tolerance, insulin sensitivity, and fat oxidation in young adults. Non-obese males and females completed fourteen 5-min sessions involving whole body passive heating at 45°C water. Changes in catecholamines, cytokines, substrate oxidation, resting energy expenditure, glucose tolerance and insulin response were assessed.

ELIGIBILITY:
Inclusion Criteria:

* healthy non-obese (BMI between 18.5 and 29.9 kg/m2) males and females;
* no diseases, or conditions that could be worsened by exposure to acute hot water and affect experimental variables;
* no participation in any excessive formal physical exercise or sports program, temperature manipulation program or exposure to extreme temperatures.

Exclusion Criteria:

* smokers;
* obesity (BMI greater than 30 kg/m2);
* needle phobia;
* taking medication and/or dietary supplements that may affect experimental variables.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in catecholamines concentration (ng/mL) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  The venous plasma adrenaline and noradrenaline concentrations (in ng/mL) were measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader
Changes in cytokines concentration (pg/mL) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  The venous serum interleukin-6 and tumor necrosis factor alpha concentrations (in pg/mL) were measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader
Change in glucose concentration (mmol/L) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  The venous glucose concentration (in mmol/L) was measured using a Glucocard X-mini plus meter.
Change in insulin concentration (μIU/mL) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  The venous serum insulin concentrations (in μIU/mL) were measured using enzyme-linked immunosorbent assay kits (Cat. No. E-EL-H2237, Elabscience, China) and a Spark multimode microplate reader (Tecan, Austria).
Change in insulin sensitivity | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Indices for insulin sensitivity/resistance assessment were computed using the homeostatic model assessment for insulin resistance, quantitative insulin-sensitivity check index (QUICKI), and the Matsuda insulin sensitivity index were calculated.
Change in substrate oxidation | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Oxygen consumption (VO2) and carbon dioxide (VCO2) output on a breath-by breath basis using a stationary MetaLyzer® 3B spiroergometry system (Cortex Biophysik GmbH) was measured at rest, and the respiratory quotient (RQ=VCO2/VO2) was computed to determine substrate utilisation.
Change in fat oxidation (g/min | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Oxygen consumption (VO2) and carbon dioxide (VCO2) output on a breath-by breath basis using a stationary MetaLyzer® 3B spiroergometry system (Cortex Biophysik GmbH) was measured at rest, and the fat oxidation (FATox; g/min) was calculated by using the equation: FATox = 1.67 × VO2 - 1.67 × VCO2,
Change in fat oxidation (g/min) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Oxygen consumption (VO2) and carbon dioxide (VCO2) output on a breath-by breath basis using a stationary MetaLyzer® 3B spiroergometry system (Cortex Biophysik GmbH) was measured at rest, and the carbohydrate oxidation (CARBox; g/min) was calculated by using the equation: CARBox = 4.55 × VCO2 - 3.21 × VO2
Change in resting energy expenditure (kcal/day) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Oxygen consumption (VO2) and carbon dioxide (VCO2) output on a breath-by breath basis using a stationary MetaLyzer® 3B spiroergometry system (Cortex Biophysik GmbH) was measured at rest, and the resting energy expenditure (REE; kcal/day) was calculated by using the Weir equation: REE = (3.941(VO2) + 1.106(VCO2)) × 1440.

SECONDARY OUTCOMES:
Change in body mass (kg) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Body mass (in kg) was evaluated using Tanita Body Composition Analyzer.
Change in fat mass (kg) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Fat mass (in kg) was evaluated using Tanita Body Composition Analyzer.
Change in fat mass (%) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Fat mass (in %) was evaluated using Tanita Body Composition Analyzer
Change in fat free mass (kg) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Fat free mass (in kg) was evaluated using Tanita Body Composition Analyzer
Change in fat free mass (%) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Fat free mass (in %) was evaluated using Tanita Body Composition Analyzer
Change in body mass index (kg/m2) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Body mass index (in kg/m2) was evaluated using Tanita Body Composition Analyzer
Change in oxygen consumption and carbon dioxide output (mL/min) | Pre-condition, post-condition (after 14 days), and after 1 month recovery
  Oxygen consumption and carbon dioxide output (in mL/min) on a breath-by breath basis using a stationary MetaLyzer® 3B spiroergometry system (Cortex Biophysik GmbH) was measured at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Brazaitis, PhD, Principal Investigator — Lithuanian Sports University
Locations (1):
- Institute of Sport Science and Innovations, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No